CLINICAL TRIAL: NCT04761029
Title: Investigation of the Efficacy of Unilateral Rhomboid Intercostal and Subserratus Plane Block Application for Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: Rhomboid Intercostal and Subserratus Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-25
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cholecystectomy; Postoperative Pain; Nerve Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grup R (Active Comparator): Unilateral Rhomboid intercostal and subserratus block + intravenous patient-controlled analgesia
  Interventions: Other: RIIS; Drug: Tramadol
- Group P (Placebo Comparator): intravenous patient-controlled analgesia
  Interventions: Drug: Tramadol

INTERVENTIONS:
Other: RIIS — unilateral Rhomboid intercostal and subserratus block
  Arms: grup R
Drug: Tramadol — intravenous patient-controlled analgesia (tramadol)

SUMMARY:
Laparoscopic surgery is frequently used today for abdominal region operations. Laparoscopy has become the preferred treatment for cholecystectomy. Patients undergoing laparoscopic cholecystectomy suffer from acute postoperative pain despite the multimodal analgesic regimen. For this type of surgery, many different field blocks have been used for postoperative analgesia.

DETAILED DESCRIPTION:
In this study, the analgesic efficacy of Unilateral Rhomboid intercostal and subserratus block was investigated in patients who had laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status I and II and who gave consent for the blocks were included in the study

Exclusion Criteria:

* bleeding disorders,
* mental incapacity,
* known allergy to the local anesthetics,
* body mass index ≥35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
tramadol consumption | Postoperative 24 hours
  tramadol consumption

SECONDARY OUTCOMES:
Numeric Rating Scale rest | postoperative 24 hours
  Numeric Rating Scale was used for pain.Pain intensity was measured using Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Numeric Rating Scale during movement | Postoperative 24 hours
  Numeric Rating Scale was used for pain.Pain intensity was measured using Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
additional analgesic use | Postoperative 24 hours
  additional analgesic use
side effect profile | Postoperative 24 hours
  side effect profile (Nausea and vomiting)
sensorial dermatomal block-level | 30 minutes after the block administration and at the postoperative 2nd hour
  Dermatomal dispersion of sensorial block to the cold stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Principal Investigator — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)